CLINICAL TRIAL: NCT05138315
Title: Quantification of Metamorphopsia Using the Alleye App Compared to the M-chart in Patients With Epiretinal Membranes a Pilot Study
Brief Title: Quantification of Metamorphopsia in Patients With Epiretinal Membranes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prof., MD, MBA, Vienna Institute for Research in Ocular Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AEM
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Alleye App and M-chart examinations will be performed pre- and postsurgically.
  Interventions: Device: Metamorphopsia quantification

INTERVENTIONS:
Device: Metamorphopsia quantification — Alleye App and M.chart examinations will be performed pre- and postsurgically.

SUMMARY:
Aim of this study is to examine metamorphopsia before and 3 months after vitrectomy with membrane peeling among patients with idiopathic epiretinal membranes. Therefore, the correlation between the Alleye App and the M-chart test before and after ERM surgery and the associations of OCT biomarkers to postsurgical changes in metamorphopsia scores will be examined.

DETAILED DESCRIPTION:
Epiretinal membranes are common disorders leading to visual loss and metamorphopsia in later stages. In most cases they are idiopathic with no identifiable cause (iERM). ERM can be visualized with optical coherence tomography (OCT) and can cause metamorphopsia, usually diagnosed with the Amsler grid or metamorphopsia chart (M-chart), which have influence on vision. ERM are surgically treated by vitrectomy and membrane peeling, however, postoperative visual acuity and quality of vision are difficult to predict. Quality of vision is highly dependent on metamorphopsia which can be an overlooked symptom. Thus, detailed examinations using M-charts prior to surgery can help to quantify the degree of metamorphopsia and might predict the potential benefit of the surgery. Recently, home monitoring tests for metamorphopsia using handheld mobile devices are becoming increasingly important. The Alleye App is one of two m-health applications with FDA approval, that is already in use for monitoring the progression of metamorphopsia in other retinal diseases such as age-related macular degeneration (AMD). It has yet to be evaluated for ERM. Aim of this study is to examine the correlation between the Alleye App and the M-chart test before and after ERM surgery and the associations of OCT biomarkers to postsurgical changes in metamorphopsia scores.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic ERM
* Sheduled surgery (vitrectomy with membrane peeling)
* Age 18 and older
* Written informed consent for participation in the study
* Metamorphopsia detected by the Amsler grid
* BCVA ≥ 0,1

Exclusion Criteria:

* Secondary ERM due to retinal tears, retinal detachment, retinal vascular diseases and uveitis
* Other macular disorders including AMD
* Previous intraocular surgery except for uncomplicated cataract surgery
* Pregnancy (pregnancy test will be performed in women of reproductive age)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Alleye App Score | 5 minutes
  The Alleye App measures the degree of metamorphopsia, the range of the Alleye App Score: 0 to 100 points, with 100 being the best achievable result, while lower values are associated with increasing degree of metamorphopsia
M-chart Scores (horizontal and vertical) | 5 minutes
  The M-charts measure the degree of horizontal and vertical metamorphopsia, the range of M-charts: 0 to 2.0, with higher values indicating a higher degree of metamorphopsia

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prof., Principal Investigator — head of department
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna, Vienna, Austria

REFERENCES:
- [Derived] Amon D, Leisser C, Schlatter A, Ruiss M, Pilwachs C, Bayer N, Huemer J, Findl O. Quantification of Metamorphopsia Using a Smartphone-Based Hyperacuity Test in Patients With Idiopathic Epiretinal Membranes: Prospective Observational Study. JMIR Perioper Med. 2025 Apr 17;8:e60959. doi: 10.2196/60959. PMID 40245427